CLINICAL TRIAL: NCT01072916
Title: The Role of Serine-Proteases in Gastrointestinal Function and Irritable Bowel Syndrome
Brief Title: Serine Proteases in Gastrointestinal Function and Irritable Bowel Syndrome (IBS)
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ian Carroll, PhD, Assistant Professor of Medicine, University of North Carolina, Chapel Hill
Other Study IDs: 08-1149; R24DK067674 (NIH)
Record Dates: First submitted 2010-02-18; First posted 2010-02-22 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2014-04

CONDITIONS: Colon, Irritable
Keywords: Colon, Irritable; Microbiota
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and Stool.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IBS: Subjects with IBS-D
- Healthy: Healthy Subjects

SUMMARY:
The proposed pilot project for this seed grant focuses on the role of intestinal serine-proteases in the pathogenesis of diarrhea-predominant IBS (D-IBS). In this study we will further assess serine-protease activity in patients with D-IBS and also explore a possible mechanism by which these proteases can lead to alterations in intestinal physiology and symptoms in these patients.

The general hypotheses for the proposed research are that (A) the levels of fecal serine-protease in patients with D-IBS are abnormally increased (B) this abnormal serine-protease activity leads to/is associated with an abnormal increase in intestinal permeability and therefore enables (C) chronic stimulation and activation of the mucosal immune system in these patients. In addition, it is aim to determine whither periodontal inflammation is associated with intestinal permeability and serine protease activity.

ELIGIBILITY:
Inclusion Criteria:

* Any sex, race, or ethnicity.
* At least 18 years of age (no upper age limit).
* D-IBS patients must meet Rome III criteria for IBS and must have been evaluated by a physician to exclude other diseases that could explain the symptoms. For the latter, patients self statement is acceptable (no official document is required).
* Participation in Dr. Whitehead's 'heterogeneity of IBS' and/or Dr. Ringel's 'intestinal inflammation in patients with D-IBS' research study.

Exclusion Criteria:

* Healthy controls must have no significant or recurring gastrointestinal symptoms.
* Patients and healthy controls should not have a serious, unstable medical condition.
* Patients and healthy controls must have had no gastrointestinal tract surgery other than appendectomy or cholecystectomy.
* Patients and healthy controls must not be pregnant (by self-report). Pregnant women will not be allowed to participate as pregnancy can affect gastrointestinal symptoms.
* Patients and healthy controls must not have a history of inflammatory bowel disease, celiac disease, or other diagnosis that could explain chronic or recurring bowel symptoms in IBS patients or controls.
* Patients and healthy controls should have no history of lactose malabsorption (by self-report).
* Patients and healthy controls should have no history of clinical symptoms of acute infections during the last 8 weeks prior to enrolment in the study.
* Patients and healthy controls should have no history of anti-inflammatory agents including aspirin, non-aspirin, non-steroid anti-inflammatory (NSAID) or steroids in the last four weeks prior to study enrollment.
* Patients should not intentionally consume probiotics or undergo antibiotic treatment during the last 4 weeks prior to enrolment in the study. If the subject consumed any of these medications, a washout period of 4 weeks will be required).
* Patients must have no history of fainting or light headedness during periods of fasting.
* Patients must not have diabetes mellitus, or any similar conditions, that would cause an adverse reaction to the sugar drink.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women of any race or ethnicity at least 18 years or older who have Diarrhea predominant Irritable Bowel Syndrome (D-IBS, n = 30) and healthy controls (n = 30).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
fecal serine protease activity | protease activity determined at at recruitment
  we will use an elisa-based method to measure the activity of serine proteases in fecal samples from IBS and HC subjects

SECONDARY OUTCOMES:
intestinal permeability | 6hrs following recruitment
  We will analyze sugar concentrations in urine to determine the level of intestinal permeability.

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Carroll, PhD, Principal Investigator — UNC Chapel Hill Department of Gastroenterology and Hepatology
Locations (1):
- University of North Carolina at Chapel Hill, Program in Digestive Health and the Department of Gastroenterology and Hepatology, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Kassinen A, Krogius-Kurikka L, Makivuokko H, Rinttila T, Paulin L, Corander J, Malinen E, Apajalahti J, Palva A. The fecal microbiota of irritable bowel syndrome patients differs significantly from that of healthy subjects. Gastroenterology. 2007 Jul;133(1):24-33. doi: 10.1053/j.gastro.2007.04.005. Epub 2007 Apr 14. PMID 17631127
- [Background] Roka R, Rosztoczy A, Leveque M, Izbeki F, Nagy F, Molnar T, Lonovics J, Garcia-Villar R, Fioramonti J, Wittmann T, Bueno L. A pilot study of fecal serine-protease activity: a pathophysiologic factor in diarrhea-predominant irritable bowel syndrome. Clin Gastroenterol Hepatol. 2007 May;5(5):550-5. doi: 10.1016/j.cgh.2006.12.004. Epub 2007 Mar 2. PMID 17336590